CLINICAL TRIAL: NCT05241613
Title: A Phase I Study to Evaluate Safety, Tolerability, PK, Pharmacodynamics, and Preliminary Anti-Tumor Activity of AC176 in Patients With Metastatic Castration Resistant Prostate Cancer Who Have Progressed on at Least Two Prior Systemic Therapies
Brief Title: A Study of AC176 for the Treatment of Metastatic Castration Resistant Prostate Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Subject benefit-risk ratio changes, sponsor decides to voluntarily terminate study
Sponsor: Accutar Biotechnology Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC176-001
Record Dates: First submitted 2022-01-17; First posted 2022-02-16 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Castration Resistant Prostate Cancer
Keywords: mCRPC; Androgen Receptor; AC176; Phase I; Androgen Receptor Degrader; First in Human
MeSH Terms: conditions — Bulbo-Spinal Atrophy, X-Linked

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AC176 Dose Escalation as Single Agent (Experimental): Single agent dose escalation of AC176. AC176 will be given orally (PO) on a 28-day cycle.
  Interventions: Drug: AC176

INTERVENTIONS:
Drug: AC176 — AC176 will be given orally (PO) on a 28-day cycle.

SUMMARY:
This clinical trial is evaluating a drug called AC176 in participants with metastatic castration resistant prostate cancer (mCRPC) who have progressed on at least two prior systemic therapies.

The main goals of this study are to:

* Identify the recommended dose of AC176 that can be given safely to participants
* Evaluate the side effects of AC176
* Evaluate pharmacokinetics of AC176
* Evaluate the effectiveness of AC176

DETAILED DESCRIPTION:
AC176-001 is a Phase I, first-in-human, open-label, multi-center dose-escalation study of AC176 given as a single agent. The AC176 is an investigational medicinal product that is a potent orally bioavailable Androgen Receptor (AR) degrader studied for the treatment of Metastatic Castration Resistant Prostate Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Males who are at least 18 years-of-age at the time of signature of the informed consent form (ICF)
2. Patients with histological, pathological, or cytological confirmed diagnosis of advanced or mCRPC who have had disease progression per Prostate Cancer Working Group 3(PCWG3) guidance following standard treatment, including approved taxane-based chemotherapy, or who are not amenable (intolerability, patient choice) to standard therapies, or for whom no therapy of proven efficacy exists.
3. Advanced or metastatic disease per PCWG3 guidance documented by either:

   • Positive bone scan (2 lesions) or metastatic lesions on computed tomography (CT)/magnetic resonance imaging (MRI) that can be followed for response.

   Or

   • Prostate-specific antigen (PSA) values with a starting value of ≥1.0 ng/mL that have increased on 3 occasions obtained a minimum of 1 week apart.
4. Patients must have progressed on at least 2 prior approved systemic therapies (in any setting), with at least 1 being abiraterone, or enzalutamide, or apalutamide or darolutamide
5. Patients who have had surgical or medical castration.
6. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 to 1
7. Life expectancy ≥3 months after the start of the treatment according to the Investigator's judgment

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from study entry:

1. Treatment with any of the following:

   * More than 2 lines of chemotherapy
   * Any systemic anti-cancer therapy, chemotherapy, biologic, or hormonal agent from a previous treatment regimen or clinical study within 4 weeks prior to the first dose of study drug. Any systemic small molecules from a previous treatment regimen or clinical study within 2 weeks or 5 half-lives (whichever is longer, not to exceed 4 weeks) prior to the first dose of study drug, except ADT for medical castration purpose.
   * Any investigational agents from a previous clinical study within 4 weeks prior to the first dose of study treatment
   * Radiation therapy (including therapeutic radioisotopes) within 4 weeks prior to first dose of study drug. Radiation for palliation within 2 weeks of study drug. Palliative radiation for the alleviation of pain due to bone metastasis will be allowed during the study
2. With the exception of alopecia and ≤ Grade 2 peripheral neuropathy, any unresolved toxicities from prior therapy greater than the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Grade 1 at the time of starting study treatment. Note: subjects with chronic Grade 2 toxicities that are asymptomatic or adequately managed with stable medication may be eligible with Sponsor approval
3. Major surgery (excluding placement of vascular access) within 4 weeks of first dose of study drug.
4. Known symptomatic brain metastases requiring steroids (above physiologic replacement doses)
5. Men who plan to father a child while in the study or within 90 days after the last administration of study treatment
6. Any condition that impairs a patient's ability to swallow whole pills. Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of AC176 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea Grade ≥2, malabsorption syndrome)
7. Any of the following cardiac criteria experienced currently or within the last 6 months:

   * Mean resting corrected QT interval (QTc) >470 msec
   * Any clinically important abnormalities (as assessed by the Investigator) in rhythm, conduction, or morphology of resting electrocardiograms (ECGs), e.g., complete left bundle branch block, third-degree heart block
   * Congestive heart failure (New York Heart Association ≥ Grade 2)
   * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years-of-age, or any concomitant medication known to prolong the QT interval
   * Left ventricular ejection fraction (LVEF) <50% or the lower limit of normal of the institutional standard.
8. As judged by the Investigator, any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, uncontrolled diabetes mellitus, active bleeding diatheses, or active infection. Screening for chronic conditions is not required. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol and/or follow-up procedures outlined in the protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male
Enrollment: 28 (Actual)
Dates: Start 2022-03-16 (Actual); Primary Completion 2024-03-05 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) from AC176 monotherapy | 28 days
  Number of subjects with DLT
Adverse events (AEs)/Serious adverse events (SAEs) | Through study completion, approximately 24 months
  Number of adverse events as characterized by type, frequency, seriousness, and relationship to AC176
Number of patients with vital signs abnormalities | Through study completion, approximately 24 months
  Vital signs abnormalities as characterized by type, frequency, severity and timing
Incidence of laboratory abnormalities as a measure of safety and tolerability of AC176 | Through study completion, approximately 24 months
  Laboratory abnormalities as characterized by type, frequency, severity and timing
Incidence of Electrocardiogram (ECG) abnormalities as a measure of safety and tolerability of AC176 | Through study completion, approximately 24 months
  Electrocardiogram (ECG) abnormalities such as heart rate, QTcF, PR, RR and QRS intervals

SECONDARY OUTCOMES:
Prostate-Specific Antigen (PSA) response rate | Throughout the study, approximately 24 months
  PSA response rate per PCWG3
Title: Duration of Response (DoR) | Throughout the study, approximately 24 months
Objective Response Rate(ORR) | Throughout the study, approximately 24 months
Time-to-Progression (TTP) | Throughout the study, approximately 24 months
Pharmacokinetic Analysis: area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC(0-inf)) | 20 weeks
Pharmacokinetic Analysis: area under the concentration-time curve over the dosing interval (AUC(0-tau)) | 20 weeks
Pharmacokinetic Analysis: maximum plasma concentration (Cmax) | 20 weeks
Pharmacokinetic Analysis: time to maximum plasma concentration (tmax) | 20 weeks
Pharmacokinetic Analysis: terminal elimination half life (t1/2) | 20 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Site 02, Denver, Colorado
  - Site 03, Sarasota, Florida
  - Site 05, Detroit, Michigan
  - Site 01, Nashville, Tennessee
  - Site 04, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/13/NCT05241613/Prot_000.pdf